CLINICAL TRIAL: NCT06366386
Title: Leveraging Existing HIV Differentiated Service Delivery Models to Screen and Treat Hypertension in Ugandan Persons Living With HIV
Brief Title: Integrating Hypertension Management in DSD for HIV
Acronym: HTN-DSD
Status: Not yet recruiting | Type: Observational
Sponsor: Infectious Diseases Research Collaboration, Uganda (Other)
Responsible Party: Sponsor
Other Study IDs: 5K43TW011963-03 (NIH)
Record Dates: First submitted 2024-03-18; First posted 2024-04-15 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Hypertension; HIV
MeSH Terms: conditions — Hypertension | interventions — Mass Screening; Seroconversion; World Health Organization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Persons living with HIV and hypertension: Persons living with HIV and hypertension aged 18 years and above will receive integrated screening (blood pressure measurement) and treatment of hypertension in their respective models of HIV care. The models of HIV care include the clinic based HIV care and community based HIV care. Treatment of hypertension will be based on a simplified one page protocol adapted from the WHO HEARTS packages for hypertension control. Health workers will be trained to titrate hypertension medications for PLHIV with hypertension using the three medications is a step wise manner: Amlodipine, Hydrochlorothiazide and Losartan.
  Interventions: Behavioral: Screening and treatment of hypertension among PLHIV in DSD models for HIV

INTERVENTIONS:
Behavioral: Screening and treatment of hypertension among PLHIV in DSD models for HIV — In all DSD models of HIV, participants will receive screening for HTN (BP measurement), treatment of hypertension using a simplified protocol of amlodipine, hydrochlorothiazide and Losartan in a stepwise manner and laboratory monitoring for HTN medication adverse events.
  Other Names: Adapted World Health Organization (WHO) HEARTS intervention for hypertension management in DSD for HIV

SUMMARY:
The goal of this implementation science study is to design evidence based and stakeholder informed implementation strategies to integrate the management of hypertension (HTN) into existing community anti-retro-viral treatment (ART) delivery models of HIV care in Uganda and evaluate their effectiveness and implementation outcomes. The main questions it aims to answer are:

1. What are the perspectives of patients (hypertensive PLHIV) on integrating hypertension care in community ART delivery models of HIV care?
2. What are the perspectives of health care providers', district leaders', and policymakers' perspectives on integrating hypertension care in community ART delivery models of HIV care?
3. What implementation strategies would support integration of the management of hypertension into existing community ART delivery models in Uganda?
4. What is the effectiveness of implementation strategies to integrate the management of hypertension care in community ART delivery models of HIV care in Uganda?
5. What are the implementation outcomes of strategies to integrate hypertension care in community ART delivery models of HIV care in Uganda?
6. What is the cumulative incidence, types and severity of HTN medication-related adverse events and their predictors among PLHIV with HTN? Investigators will use qualitative research methods to explore key stakeholders' perspectives and preferences on integrating hypertension care in community ART delivery models in Uganda; design implementation strategies that integrate the management of hypertension into existing community ART delivery models; determine the effectiveness of implementation strategies that integrate the management of hypertension in community ART delivery models; evaluate implementation outcomes of strategies that integrate hypertension care in community ART delivery models; determine the cumulative incidence, types and severity of medication-related adverse events and their predictors; and assess the patients and provider costs, health related quality of life, cost-effectiveness of leveraging existing HIV differentiated service delivery models to screen and treat HTN among persons with HIV in Uganda.

DETAILED DESCRIPTION:
Introduction: Over a billion people worldwide have hypertension (HTN), although 46% are unaware. Approximately a third of adult people living with HIV (PLHIV) have hypertension (HTN), partly due to increased longevity, HIV related inflammation and antiretroviral therapy (ART) use. The high prevalence of HTN exposes PLHIV to an increased risk of ischemic heart disease, stroke and kidney disease. Community delivery of antiretroviral therapy (ART) improves retention and viral load suppression for PLHIV. However, HTN management is not yet integrated into community ART delivery models in which over 50% of PLHIV receive care because initial integration efforts are focused at health facilities. Additionally, the proportion of hypertensive PLHIV with controlled blood pressure is still low (5%) in Uganda. Thus, integrating the management of HTN into community ART models could improve HTN control in PLHIV and reduce the cardiovascular diseases (CVD) risk. Treating HIV, HTN and other non-communicable diseases (NCDs) concurrently raises concerns for medication-related adverse events, including but not limited to: adverse signs and symptoms (cough, angioedema, peripheral edema) and laboratory abnormalities (hypo-/hyper-kalemia, hyponatremia, hyperglycemia, hyperlipidemia). Yet, little is known about the burden and profile of such adverse events among patients concurrently treated for HIV and HTN in low-income countries like Uganda. Availability of such information is likely to improve the safety and acceptability of integrated HIV-HTN care.

Aims: This study aims: 1) To explore key stakeholders' perspectives and preferences on integrating hypertension care in community ART delivery models in Uganda; 2) To design implementation strategies that integrate the management of hypertension into existing community ART delivery models; 3) To determine the effectiveness of implementation strategies that integrate the management of hypertension in community ART delivery models and 4) To evaluate implementation outcomes of strategies that integrate hypertension care in community ART delivery models, 5) To determine the cumulative incidence, types and severity of medication-related adverse events and their predictors 6) To assess the patients and provider costs, health related quality of life, cost-effectiveness of leveraging existing HIV differentiated service delivery models to screen and treat HTN among persons with HIV in Uganda.

Methods: Investigators will use mixed methods research to conduct a formative study to explore stakeholders' perspectives and preferences of integrating HTN care into community ART delivery models. Using the Consolidated Framework for Implementation Research (CFIR), investigators will determine factors that influence the integration of HTN management into community ART models. Investigators will then design implementation strategies to integrate HTN management into community ART models using group model building. Investigators will do this through rigorous engagement of stakeholders who participate in the implementation of HIV and HTN services. These will include healthcare providers, health leaders at district and health facilities as well as patient representatives. To develop generalizable implementation strategies, investigators will use the widely validated CFIR-Expert Recommendations to Implement Change (CFIR-ERIC) tool to classify the strategies. Investigators will then name, define and operationalize the implementation strategies according to Proctor et al. Then, investigators will implement and determine effectiveness of the implementation strategies using an interrupted time series analysis (ITSA) across four health facilities and their community ART delivery models. in addition, investigators will leverage a cohort of ageing PLHIV receiving both HIV and HTN care to conduct baseline laboratory investigations, with a repeat of these tests at intervals of one and six months post initiation of HTN medicines, to profile adverse events associated with HTN medications among these PLHIV. Finally, investigators will evaluate the implementation and process outcomes of the implementation strategies. Investigators will do this by quantifying HIV and HTN indicators and qualitatively exploring stakeholders' barriers and facilitators towards the integrated management of HTN within community ART models. Investigators will use the Reach Effectiveness Adoption Implementation and Maintenance (RE-AIM) framework of implementation science to conduct the process evaluation.

Implications of the proposed research: This study will use rigorous implementation science methods to design implementation strategies and determine their effectiveness in integrating HTN management into community-based ART delivery models. The implementation strategies may lead to improved dual control of HIV and HTN in patients who receive care in the community. By profiling HTN medication-related adverse events and their predictors among an ageing HIV population, our study will provide a benchmark for such events, as well as build capacity on monitoring and managing medication-related adverse events among PLHIV with HTN and other NCDs. Our theory of change for integrating HTN management into community-based ART delivery models will inform Ugandan HIV and HTN guidelines and could be generalizable to other low income settings. Study findings will also demonstrate the utility of implementation science in the chronic care of HTN and HIV in the community.

ELIGIBILITY:
Inclusion Criteria:

* Adult PLHIV receiving HIV care either through clinic or community based ART delivery at the selected health facilities.

Exclusion Criteria:

* This study will be implemented in the real world setting and the proposed HTN medications are already authorized for use in Uganda. Therefore, we will not exclude any patient from accessing HTN services (screening, treatment and monitoring) unless if any patients decline taking the medicines for whichever reason. However, special patient categories including pregnant mothers, diabetic patients and those with kidney or heart disease will be referred for specialized care.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will include all adult PLHIV receiving HIV care either through clinic or community based ART delivery at the selected health facilities. In this controlled pre-post study, all PLHIV receiving care will be targeted to receive HTN care which will include screening, treatment and monitoring
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Number of PLHIV with controlled blood pressure (both systolic and diastolic blood pressure) | Six months after starting treatment of hypertension
  Number of PLHIV with HTN who will achieve Blood pressure control (both systolic and diastolic blood pressure) after starting treatment.
% of PLHIV with controlled blood pressure (both systolic and diastolic blood pressure) | Six months after starting treatment of hypertension
  Proportion of PLHIV with HTN who will achieve Blood pressure control (both systolic and diastolic blood pressure) after starting

SECONDARY OUTCOMES:
Mean blood pressure (both systolic and diastolic blood pressure) | 12 months after starting treatment
  Mean blood pressure (both systolic and diastolic blood pressure) of the study participants
Number and % of hypertensive PLHIV with suppressed Viral load | 12 months after starting treatment
  Number and proportion of hypertensive PLHIV with suppressed Viral load
Number and % of patients retained in care | 12 months after starting treatment
  Number and proportion of patients retained in care and number
Number and % of PLHIV screened for HTN at least once in six months | 12 months after starting treatment
  Number and proportion of PLHIV screened for HTN at least once in six months
Implementation costs | 12 months after starting treatment
  Cost of implementing strategies to integrate the management of hypertension into differentiated service delivery for HIV.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Muddu, MMED, Principal Investigator — Infectious Diseases Research Collaboration, Uganda
Locations (1):
- Infectious Diseases Research Collaborations (IDRCUganda), Kampala, Central Region, Uganda

IPD SHARING:
Plan to Share IPD: No
We will not share individual participant data (IPD) with other researchers outside the Infectious Diseases Research Collaboration (IDRC).